CLINICAL TRIAL: NCT04326959
Title: Implantation of Mesenchymal Stem Cell, Conditioned Medium, or Triamcinolone Acetonide for Keloid Regression: Immunohistochemistry, Histopathology and Imaging Study
Brief Title: Implantation of Mesenchymal Stem Cell, Conditioned Medium, or Triamcinolone Acetonide for Keloid
Acronym: Keloid
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/KLD/03/2020
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Keloid
Keywords: Keloid; Allogeneic Mesenchymal Stem Cells; Umbilical Cord; Conditioned Medium
MeSH Terms: conditions — Keloid | interventions — Culture Media, Conditioned; Secretome; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- UC-MSCs + CM (Experimental): A patient will be given UC-MSCs 2 million cells / cm3. After 3 weeks, the patient will be given CM 1 cc / cm3. The maximum size of Keloid is 15 cm per patient.
  Interventions: Biological: Umbilical Cord-Mesenchymal Stem Cells and Conditioned Medium; Biological: Conditioned Medium
- CM + CM (Experimental): A patient will be given CM 1 cc / cm3. After 3 weeks, the patient will be given CM 1 cc / cm3. The maximum size of Keloid is 15 cm per patient.
  Interventions: Biological: Conditioned Medium
- Triamcinolon acetonide (Experimental): A patient will be given Triamcinolone acetonide 40 mg / cc / cm3. After 3 weeks the patient will be given Triamcinolone acetonide 40 mg/cc / cm3. The maximum size of Keloid is 15 cm per patient.
  Interventions: Biological: Triamcinolone Acetonide

INTERVENTIONS:
Biological: Umbilical Cord-Mesenchymal Stem Cells and Conditioned Medium — Injection of Allogeneic Umbilical Cord Mesenchymal Stem Cells 2 million cell/cm3 in Nacl 1 cc/million cell and booster with Conditioned Medium 1 cc/cm3 in 3 weeks later. All treatment via intralesional injection. The maximum size of the keloid is 15 cm.
  Arms: UC-MSCs + CM
Biological: Conditioned Medium — Injection of Conditioned Medium 1 cc/cm3 and booster with Conditioned Medium 1 cc/cm3 in 3 weeks later. All treatment via intralesional injection. The maximum size of the keloid is 15 cm.
  Other Names: Secretome
  Arms: CM + CM; UC-MSCs + CM
Biological: Triamcinolone Acetonide — Injection of Triamcinolone Acetonide 40 mg/cc/cm3 and booster in 3 weeks later. All treatment via intralesional injection. The maximum size of the keloid is 15 cm.
  Arms: Triamcinolon acetonide

SUMMARY:
The clinical trial will be carried out at the Gatot Soebroto Army Central Hospital, Jakarta and planned from June 2020 to December 2020. Clinical trials of Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs) and Conditioned Medium Umbilical Cord-Mesenchymal Stem Cells (CM UC-MSCs) for Keloid were designed in three groups. Group 1 injected with The UC-MSCs at a dose of 2 million cells / cm3 using a 1 cc injection syringe (27G) by intra-lesion injection and booster with CM UC-MSCs at a dose of 1 cc / cm3 using a 1 cc injection syringe (27G) by intra-lesion injection and booster with CM UC-MSCs at the same dose 3 weeks later. Group 3 injected with Triamcinolon acetonide (TA) at a dose of 40 mg / cc / cm3 using 1 cc (27 G) syringe and booster with TA at 3 weeks later. The study subjects each group amounted to 7 patients suffering from Keloid. Patients were evaluated for 3 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Surgery history of more than 3 months
* Has keloid that the maximum size is 15 cm and thickness is 3-5 mm

Exclusion Criteria:

* Patients with kidney failure
* Pregnancy
* Breastfeeding
* Liver dysfunction
* Blood disorders
* Currently receiving immunosuppressant therapy (chemotherapy or steroids)
* Refusing to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-08 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Alfa SMA-1 | 3 month after injection
  Biomarker
Collagen type 1 | 3 moth after injection
  Biomarker

SECONDARY OUTCOMES:
Core Biopsy/Histopathology | 3 month after injection
  Too evaluate histology of keloid
Ultrasonography | 3 month after injection
  To see image inside the body